CLINICAL TRIAL: NCT06478563
Title: Investigating the Exposure of NNC0487-0111 in Different Oral Formulations and the Effect of Food Intake on Pharmacokinetics of NNC0487-0111 in Participants With Overweight or Obesity
Brief Title: A Research Study Looking at Different Oral Formulations and the Effect of Food Intake on How the Medicine NNC0487-0111 Behaves in the Body of Participants Living With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NN9487-7980; U1111-1300-3720 (Other: Universal Trial Number)
Record Dates: First submitted 2024-06-24; First posted 2024-06-27 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single-blinded to the investigator (to the formulation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase A: NNC0487-0111 (formulation D) (Experimental): Participants will receive once daily dose of six different dose levels (1-6) of NNC0487-0111 (formulation D) at increasing doses (the dose will be escalated every 3 weeks).
  Interventions: Drug: NNC0487-0111 (formulation D)
- Phase A: NNC0487-0111 (formulation C) (Active Comparator): Participants will receive once daily dose of six different dose levels (1-6) of NNC0487-0111 (formulation C) at increasing doses (the dose will be escalated every 3 weeks).
  Interventions: Drug: NNC0487-0111 (formulation C)
- Phase B: NNC0487-0111 (formulation D) (Experimental): Participants will receive once daily dose of dose level 6 of NNC0487-0111 (formulation D).
  Interventions: Drug: NNC0487-0111 (formulation D)
- Phase B: NNC0487-0111 (formulation C) (Active Comparator): Participants will receive once daily dose of dose level 6 of NNC0487-0111 (formulation C).
  Interventions: Drug: NNC0487-0111 (formulation C)

INTERVENTIONS:
Drug: NNC0487-0111 (formulation D) — Participants will receive NNC0487-0111 (formulation D) tablet once daily.
  Arms: Phase A: NNC0487-0111 (formulation D); Phase B: NNC0487-0111 (formulation D)
Drug: NNC0487-0111 (formulation C) — Participants will receive NNC0487-0111 (formulation C) tablet once daily.
  Arms: Phase A: NNC0487-0111 (formulation C); Phase B: NNC0487-0111 (formulation C)

SUMMARY:
This study consists of two phases: Phase A and Phase B. Participants are being asked to participate in both phases. Phase A of this study is comparing two formulations of a study medicine called NNC0487-0111 for weight control in people with overweight or obesity. Phase B of this study is testing how taking NNC0487-0111 at the same time as a meal affects the way NNC0487-0111 works in participants body. The aim of this study is to compare how two different formulations of NNC0487-0111 behave in the body, and how their function is affected when they are taken with or without a meal. Participants will either get NNC0487-0111 Formulation C, or NNC0487-0111 Formulation D. Both formulations are given as tablets. Which treatment participants get is decided by chance. Oral NNC0487-0111 is a new medicine which cannot be prescribed by doctors but has previously been tested in humans. The study will last for about 5 - 6 months (155-184 days).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-64 years (both inclusive)
* Body mass index (BMI) between 27.0 and 39.9 kilogram per meter square (kg/m^2) (both inclusive)
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
* Any laboratory safety parameters at screening outside the below laboratory ranges, see designated reference range documents for specific values:
* Vitamin D (25-hydroxycholecalciferol) less than (<) 12 ng/mL (30 Nanometer (nM)) at screening
* Parathyroid hormone (PTH) outside normal range at screening
* Total calcium outside normal range at screening
* Calcitonin greater than or equal to (≥) 50 pg/mL at screening
* Amylase greater than or equal to (≥) 2 times upper limit of normal
* Lipase greater than or equal to (≥) 2 times upper limit of normal
* Glycated hemoglobin (HbA1c) greater than or equal to (≥) 6.5 % (48 millimoles per mole (mmol/mol)) at screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Phase A: The area under the NNC0487-0111 plasma concentration-time curve during a dosing interval at steady state | From pre-dose to after dosing on days 21, 42, 63, 84, 105 and 126
  Measured as hours*nanomoles per liter (h*nmol/L)

SECONDARY OUTCOMES:
Phase A: The maximum observed plasma concentration of NNC0487-0111 at steady state | From pre-dose to after dosing on days 21, 42, 63, 84, 105 and 126
  Measured as nanomoles per liter (nmol/L)
Phase A: The time from dose administration to maximum observed plasma concentration of NNC0487-0111 at steady state | From pre-dose to after dosing on days 21, 42, 63, 84, 105 and 126
  Measured as hours
Phase B: The area under the NNC0487-0111 plasma concentration-time curve | From pre-dose to after dosing on day 132
  Measured as h*nmol/L
Phase B: The maximum plasma concentration of NNC0487-0111 after the last dose | From pre-dose to after dosing on day 132
  Measured as nmol/L
Phase B: The time to maximum observed plasma concentration of NNC0487-0111 after the last dose | From pre-dose to after dosing on day 132
  Measured as hours
Phase B:The terminal half-life of NNC0487-0111 after the last dose | From pre-dose on day 132 until completion of the end of study visit (day 153)
  Measured as hours
Number of treatment emergent adverse events (TEAE) | From time of trial product administration (Visit 2, day 1) until completion of the end of study visit (day 153)
  Measured as number of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Celerion, Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com